CLINICAL TRIAL: NCT06806267
Title: Study of the Effectiveness of Virtual Exposure Therapy (VRET) in Combination With Transcranial Direct Current Stimulation (tDCS) in the Treatment of Veterans and Civilians With PTSD in Wartime Ukraine
Brief Title: Study of the Effectiveness of VRET Combined With tDCS in the Treatment of PTSD in Ukrainian Veterans and Civilians
Acronym: AVRE-U
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Malek Bajbouj (Other)
Collaborators: Bogomolets National Medical University (Other); Khmelnytsky Regional Institution for psychiatric care (Unknown); Ternopil Regional Clinical Psychoneurological Hospital (Unknown); Danylo Halytsky Lviv National Medical University (Other); Dnipropetrovsk Clinical Multidisciplinary Hospital for Psychiatric Care (Unknown); Clinical Hospital 'Psychiatry' of the executive body of the Kyiv City Council (Unknown)
Responsible Party: Sponsor-Investigator, Malek Bajbouj, Prof. Dr. med., Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 314159265358979323846264338
Record Dates: First submitted 2025-01-16; First posted 2025-02-04 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: PTSD - Post Traumatic Stress Disorder
Keywords: PTSD; VRET; tDCS; Virtual Reality; Exposure therapy; Veterans; Ukraine
MeSH Terms: conditions — Combat Disorders; Stress Disorders, Post-Traumatic | interventions — Transcranial Direct Current Stimulation; Implosive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- VRET (Experimental): Participants will receive Virtual reality exposure therapy
  Interventions: Device: Virtual reality exposure therapy
- VRET an tDCS (Experimental): Participants will receive Virtual reality exposure therapy and transcranial direct current stimulation
  Interventions: Device: Virtual reality exposure therapy; Device: transcranial direct current stimulation
- Treatment as usual (Active Comparator): Participants will receive non-virtual reality exposure therapy
  Interventions: Behavioral: Imaginal exposure therapy

INTERVENTIONS:
Device: Virtual reality exposure therapy — Exposure therapy applied through virtual reality goggles, controlled by a clinician
  Arms: VRET; VRET an tDCS
Device: transcranial direct current stimulation — transcranial direct current stimulation applied to the vmpfc, 2mA
  Arms: VRET an tDCS
Behavioral: Imaginal exposure therapy — Imaginal exposure therapy
  Arms: Treatment as usual

SUMMARY:
A new method is being tested to assist individuals in Ukraine with Post-Traumatic Stress Disorder (PTSD), including veterans and civilians affected by war. The study is a collaboration among Ukrainian healthcare institutions and the Charité Berlin.

What is PTSD?

PTSD can occur after a distressing or traumatic experience, such as exposure to war. It can result in persistent negative memories, nightmares, heightened nervousness, or avoidance of reminders associated with the event.

Purpose of the Study

Two innovative treatments for PTSD are being tested:

1. Virtual Reality Therapy: This approach uses specialized goggles to create a safe and realistic virtual environment where individuals can confront memories and process emotions with guidance from a therapist.
2. Brain Stimulation Therapy (tDCS): This method applies a gentle electrical current to the scalp to support improved emotional regulation by the brain.

The study aims to determine whether combining these two treatments is more effective than using virtual reality therapy alone.

Participant Involvement

Participants will:

* Attend 10 therapy sessions over several weeks.
* Use virtual reality goggles to engage with safe scenarios related to their memories, guided by a therapist.
* Potentially receive brain stimulation therapy during some virtual reality sessions.
* Learn relaxation techniques to help manage stress and enhance emotional control.

Potential Benefits for Participants

* These treatments may reduce symptoms such as intrusive memories, anxiety, and depression.
* Participants may experience increased calmness, resilience, and improved ability to manage daily life.

This study also has the potential to advance PTSD treatment methods for others in the future.

DETAILED DESCRIPTION:
This research initiative, supported by Charité - Universitätsmedizin Berlin, involves collaboration among six Ukrainian institutions to investigate the effectiveness of Virtual Reality Exposure Therapy (VRET) combined with Transcranial Direct Current Stimulation (tDCS) for the treatment of PTSD in war veterans and civilians.

Background and Rationale

Reports since 2015 indicate that approximately 27.7% of individuals involved in the Anti-Terrorist Operation (ATO) in Ukraine have been diagnosed with PTSD, highlighting a critical need for innovative treatments.

Exposure therapy is a well-established treatment for PTSD, helping individuals process traumatic memories through techniques such as gradual exposure and arousal control. However, traditional approaches often result in high dropout rates due to the emotional intensity required. Virtual Reality Exposure Therapy (VRET) offers a promising alternative by providing immersive, interactive, and controlled environments that facilitate emotional processing and reduce avoidance behaviors. A culturally adapted Ukrainian version of the VRET protocol, developed in 2024 at the Bogomolets National Medical University, has shown potential for addressing trauma-specific needs in Ukrainian PTSD patients.

tDCS is a non-invasive neuromodulation technique that applies low electrical currents to the scalp to influence brain activity. It has shown promise in alleviating PTSD-related symptoms such as anxiety, depression, and emotional dysregulation. Combining tDCS with VRET may enhance treatment outcomes by leveraging neuroplasticity to improve emotional regulation and cognitive processing.

This study aims to validate a culturally adapted VRET protocol for PTSD treatment in Ukraine and evaluate whether combining it with tDCS further enhances therapeutic outcomes.

Treatment Protocols

Virtual Reality Exposure Therapy (VRET)

The VRET protocol involves ten 60-minute sessions structured in two phases:

* Phase 1: Screening, informed consent, and baseline assessments.
* Phase 2 (Sessions 1-10): Gradual exposure to trauma-related virtual environments with guided psychological interventions, including psychoeducation, relaxation techniques, and cognitive restructuring. Sessions are tailored to individual needs with real-time adjustments by therapists.

Session Highlights:

* Session 1: Psychoeducation about PTSD and relaxation training.
* Sessions 3-5: Gradual introduction of tailored VR scenarios with controlled activation of traumatic memories.
* Sessions 6-9: Narrative construction of traumatic experiences, with continued relaxation and emotional regulation techniques.
* Session 10: Assessment of emotional state and development of self-stabilization skills for daily life.

tDCS-Augmented VRET (tDCS-VRET) The tDCS-VRET protocol incorporates tDCS during VRET sessions to enhance neuromodulation. Sessions are identical to the VRET protocol, with the addition of tDCS targeting the dorsolateral prefrontal cortex.

* tDCS Parameters: 2 mA current, with 30-second ramp-up and ramp-down phases, not exceeding 30 minutes per session.
* Sessions include tDCS alongside VR exposure scenarios, relaxation techniques, and physiological monitoring to reinforce adaptive coping.

Technical Specifications

* VRET Equipment: Oculus Quest 2 headset with Unity3D-based VR software by "VR Mentality" LLC, enabling real-time therapist adjustments and personalized trauma-related scenarios.
* tDCS Equipment: NeuroFlow device with app-controlled interface, silicone electrodes, and 2 mA current capacity.

Objectives

* Assess the effectiveness of culturally adapted VRET for PTSD in Ukrainian patients.
* Evaluate the added benefit of tDCS in enhancing VRET outcomes, including reductions in PTSD symptoms, anxiety, and depression, and improvements in emotional regulation and quality of life.

This protocol offers an innovative and integrative approach to PTSD treatment by combining state-of-the-art virtual reality technology with neuromodulation to address the specific needs of Ukrainian trauma survivors.

ELIGIBILITY:
Inclusion Criteria:

* Participants are eligible to be included in the study only if all of the following criteria apply:

Age · The participant is 18 to 75 years of age, inclusive, at the time the informed consent form (ICF) is signed.

Type of Participant and Disease Characteristics:

* The participant has a current diagnosis of PTSD as defined by the CAPS-5, with a CAPS-5 Total Symptom Severity Score of ≥30 at the Screening Visit and Baseline Visit and no >25% change in score from Screening to Baseline.
* The participant's index trauma event must have occurred when the participant was ≥13 years of age.

  1. In the opinion of the Investigator the participant has a high probability for adherence with and completion of the study.
  2. The participant has the ability to comply with study procedures.
  3. The participant is fluent in Ukrainian and able to understand and comply with written and verbal protocol-related requirements.
  4. The participant has received study inclusion approval through an adjudication process as to final suitability for the study.

Exclusion Criteria:

1. Individuals with Epilepsy, Seizures or Severe Brain Injuries
2. Individuals with Implanted Electronic Devices (Pacemakers, Cochlear Implants, etc.)
3. Individuals with Scalp or Skin Issues at electrode placement sites
4. Pregnant Individuals
5. Individuals with tinnitus

Medical Conditions

1. It has been less than 6 months since the participant's index trauma event occurred, at the time of the Screening Visit.
2. The participant has current and ongoing exposure to the trauma that caused their PTSD.
3. The participant has complex PTSD, defined as a condition that may develop following exposure to an event or series of events of an extreme and prolonged or repetitive nature, which the participant experienced as extremely threatening or horrific and from which escape was difficult or impossible (e.g., torture, slavery, genocide campaigns, prolonged domestic violence, repeated childhood sexual or physical abuse). If affect dysregulation and interpersonal dysfunction are primary over other core PTSD symptoms, in the Investigator's opinion, participants should be excluded.
4. The participant has severe depression as measured by a score of ≥35 on the Montgomery-Åsberg Depression Rating Scale (MADRS) at the Screening Visit.
5. The participant has bipolar disorder, borderline personality disorder and other psychotic disorders as identified at the Screening Visit using the Structured Clinical Interview for DSM-5 Disorders - Clinical Trials Version (SCID-5-CT) and Personality Disorders (SCID-5-PD).
6. The participant has a history of moderate to severe traumatic brain injury.
7. The participant has a history of seizure disorders, uncontrolled sleep apnea or severe neurologic disease.
8. The participant has any moderate or severe substance use disorder according to DSM-5 in the 12 months prior to the Screening Visit.
9. The participant has a score of >15 points on the Alcohol Use Disorders Identification Test (AUDIT) at the Screening Visit.
10. The participant is at an increased risk of suicide, defined as:

    * Any suicide attempt in the 12 months prior to the Screening Visit disclosed by the participant using the Columbia Suicide Severity Rating Scale (C-SSRS)
    * Any suicidal ideation with intent (yes to item 4 and/or 5) in the past 6 months or suicidal behaviour in the past 12 months, as captured at the Screening Visit or Baseline Visit using the C-SSRS
    * A score >4 on item 10 of the MADRS at the Screening Visit.
11. The participant has a systolic blood pressure value >140 mmHg or diastolic blood pressure value >90 mmHg at the Screening Visit or Baseline Visit. Two repeat measures are allowed at the discretion of the Investigator.
12. The participant has negative experience or reaction to VR technology.
13. The participant has significant cognitive impairments affecting instruction comprehension.
14. The participant has any clinically significant ECG abnormality as determined by the Investigator at the Screening Visit.
15. The participant has pronounced adverse physiological reactions to VR that remain unmanageable
16. The participant is receiving concurrent trauma-based psychotherapy such as Cognitive Behaviour Therapy, Prolonged Exposure Therapy, Eye Movement Desensitization and Reprocessing Therapy.

Prior/Concomitant Therapy

1. The participant is receiving concurrent trauma-based psychotherapy such as Cognitive Behaviour Therapy, Prolonged Exposure Therapy, Eye Movement Desensitization and Reprocessing Therapy.
2. The participant has used marijuana or cannabinoid containing products daily (occasional use is allowed) for recreational use or self-medication (prescribed or otherwise) for the treatment of symptoms of PTSD or any other CNS disorder within 60 days of the Screening Visit.

Prior/Concurrent Clinical Study Experience

1. The participant is currently enrolled in OR has previously participated in another investigational study in which an investigational medication (e.g., drug, vaccine, invasive device) was administered within 30 days before the ICF for this study is signed.

Other Exclusions

1. The participant is a member of the Ukrainian military currently serving on active duty.
2. The participant is in the process of litigating for compensation for a psychiatric disorder. Participants who are in the process of applying for medical or Veterans Affairs benefits and/or those who have settled a disability claim prior to enrolment in the trial are eligible.
3. The participant is not suitable to participate in the study, in the opinion of the investigator, because of clinically significant findings on medical history that could interfere with the objectives of the study or put the participant at risk or for any other reason the investigator deems applicable.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 514 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
PTSD Symptoms | Before treatment until after treatment as well as 3-month and 6-month follow ups
  CAPS-5 (Clinician-Administered PTSD Scale for DSM-5)
  * Minimum Value: 0
  * Maximum Value: 80
  * Higher Scores: Indicate worse outcomes, reflecting more severe PTSD symptoms.
PTSD Symptoms as measured by PCL-5 | Before treatment until after treatment as well as 3-month and 6-month follow ups
  PCL-5 (Posttraumatic Stress Disorder Checklist for DSM-5)
  * Minimum Value: 0
  * Maximum Value: 80
  * Higher Scores: Indicate worse outcomes, as they reflect more severe PTSD symptoms.

SECONDARY OUTCOMES:
Symptoms of depression | Before and after end of treatment as well as at 3-month and 6-month follow ups
  MADRS (Montgomery-Åsberg Depression Rating Scale)
  * Minimum Value: 0
  * Maximum Value: 60
  * Higher Scores: Indicate worse outcomes, reflecting more severe depression symptoms.
Quality of life | Before and after end of treatment as well as at 3-month and 6-month follow ups
  SF-36 (36-Item Short Form Health Survey)
  * Minimum Value: 0
  * Maximum Value: 100
  * Higher Scores: Indicate better outcomes, reflecting better health-related quality of life.
Framework of acceptability Questionnaire | Before and after end of treatment as well as at 3-month and 6-month follow ups
  Framework of acceptability Questionnaire
  * Minimum Value: 0
  * Maximum Value: 40
  * Higher Scores: Indicate better outcomes, reflecting higher levels of acceptability of the Intervention .
Suicidal Ideation | Before and after end of treatment as well as at 3-month and 6-month follow ups
  C-SSRS (Columbia-Suicide Severity Rating Scale)
  * Minimum Value: 0 (No suicidality)
  * Maximum Value: 25
  * Higher Scores: Indicate worse outcomes, reflecting increased severity of suicidal ideation or behavior.
Anxiety | Before and after end of treatment as well as at 3-month and 6-month follow ups
  GAD-7 (Generalized Anxiety Disorder-7)
  * Minimum Value: 0
  * Maximum Value: 21
  * Higher Scores: Indicate worse outcomes, reflecting higher levels of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Malek Bajbouj, Prof. Dr. med, Principal Investigator — Charité

IPD SHARING:
Plan to Share IPD: Yes
to be decided